CLINICAL TRIAL: NCT05800418
Title: Phase I Clinical Study of Single-center, Randomized, Double-blind, Single-dose, Parallel Comparison of the Pharmacokinetics and Safety of Ramucirumab Injection and Cyramza® in Healthy Male Volunteers
Brief Title: Clinical Study to Compare the Pharmacokinetics and Safety of Ramucirumab Injection With Cyramza ® in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZDTQ-2019-LMLDK
Record Dates: First submitted 2023-03-24; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2019-10

CONDITIONS: Gastric Cancer; Non-small Cell Lung Cancer; Colo-rectal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms | interventions — Ramucirumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ramucirumab injection (Experimental): 8mg/kg, Single intravenous infusion
  Interventions: Drug: Ramucirumab Injection
- Cyramza (Active Comparator): 8mg/kg, Single intravenous infusion
  Interventions: Drug: Ramucirumab Injection [Cyramza]

INTERVENTIONS:
Drug: Ramucirumab Injection — Ramucirumab injection biosimilar products manufactured by Chia Tai Tianqing Pharmaceutical,
  Arms: Ramucirumab injection
Drug: Ramucirumab Injection [Cyramza] — Ramucirumab Injection is a humanized monoclonal antibody based on the human immunoglobulin G1(IgG1) skeleton sequence, developed by Eli Lilly Co., the bran name is Cyramza. Ramucirumab is a vascular endothelial growth factor receptor 2 (VEGFR2) antagonist that specifically binds to VEGF receptor 2 and blocks VEGFR ligand, VEGF-A, VEGF-C, and VEGF-D binding to the receptor. As a result, Ramucirumab inhibits ligand-stimulated VEGF receptor 2 activation, thereby inhibiting ligand-induced proliferation, and human endothelial cell migration. Ramucirumab inhibits angiogenesis, thereby blocking the tumor's blood vessel supply.
  Arms: Cyramza

SUMMARY:
Ramucirumab is a biosimilar drug of CYRAMZA® produced by Chiatai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., LTD. It is a vascular endothelial growth factor receptor 2 (VEGFR-2) antagonist. This single-center, randomized, double-blind, single-dose, parallel phase I study of Ramucirumab injection versus Cyramza ® in healthy male volunteers was designed to evaluate the similarities in pharmacokinetics, tolerance, safety and immunogenicity of Ramucirumab and CYRAMZA®.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent form before the study and fully understand the study content, process and possible adverse reactions;
* Be able to complete the study according to the requirements of the test plan;
* Male subjects aged 18-65 years (included);
* The subject should weigh at least 50kg. Body mass index (BMI) = weight (kg)/ height2(m2), BMI in the range of 19 to 26 (included);
* Health status: no mental abnormality, no medical history of abnormal cardiovascular system, nervous system, respiratory system, digestive system, urinary system, endocrine system and metabolism;
* Normal or abnormal vital signs, physical examination, laboratory examination, electrocardiogram and imaging examination with no clinical significance;
* Have no pregnancy plan and voluntarily take effective contraception measures from 2 weeks before the study drug administration to at least 6 months after the last dose.

Exclusion Criteria:

* Have a history of neuropsychiatric system, respiratory system, cardiovascular system, digestive system, hemolymph system, liver and kidney insufficiency, endocrine system, skeletal and musculoskeletal system disease or other diseases, and the investigators judge that this history may affect drug metabolism or safety;
* Known allergic to Ramucirumab or its excipients; Known history of allergic diseases or allergic constitution;
* History of hypertension or abnormal blood pressure at screening/baseline measurement (systolic blood pressure (SBP) > 140 mmHg, and/or diastolic blood pressure (DBP) >90 mmHg, confirmed by one repeat measurement on the same day);
* A history of clinically significant albuminuria (urine routine examination, albuminuria 2+ and above) or albuminuria as assessed by the investigator;
* Had received treatment of Ramucirumab or VEGFR2 receptor antagonist, or other antibody or protein drugs that target VEGFR2 receptor;
* Had received any live viral vaccine within 2 months prior to study drug infusion, or required vaccination between the screening period and the end of the study, had used any monoclonal antibody or biologic drug within 12 months prior to study drug administration, or planned to receive any monoclonal antibody or biologic drug within 12 months after study drug administration;
* had unhealed wound ulcers or fractures, or had undergone major surgery within 3 months prior to study drug infusion or expected to undergo major surgery during the study period or within 2 months after study completion;
* had taken any prescription drugs, over-the-counter drugs, any vitamin products, or herbs within 14 days prior to use of the study drug;
* Patients with abnormal examinations and clinical significance during the screening period;
* Blood donation or significant blood loss within 3 months prior to use of the study drug (>450 mL);
* Have taken the study drug or participated in any clinical trial of the drug within 3 months prior to the use of the study drug;
* Smokers who smoked more than 5 cigarettes a day in the 3 months before the test;
* Test positive for alcohol or have a history of alcohol abuse (14 units of alcohol per week: 1 unit =360 mL of beer or 45 mL of 40% spirits or 150 mL of wine);
* Test positive for drugs or have a history of drug abuse in the past five years or have used drugs in the three months prior to the test;
* Hepatitis (including hepatitis B and C), AIDS, syphilis positive screening;
* Patients with difficulty in venous blood collection or who cannot tolerate venipuncture;
* Unable or unable to comply with ward management regulations, poor compliance during the study, or unable to follow protocol requirements to complete the study;
* Subjects unable to complete the experiment due to personal reasons;
* Conditions considered unsuitable for inclusion by other researchers.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Area under drug concentration - time curve (AUC0-t) | Within 60 minutes before administration to 1680 hours after administration.
  Area under the curve from zero to the lowest detectable blood drug concentration.

SECONDARY OUTCOMES:
Area under drug concentration - time curve (AUC0-∞) | Within 60 minutes before administration to 1680 hours after administration.
  The area under the curve extrapolating from zero to infinity.
Peak concentration (Cmax) | Within 60 minutes before administration to 1680 hours after administration.
  Peak maximum plasma drug concentration
Peak concentration time (Tmax) | Within 60 minutes before administration to 1680 hours after administration.
  Time to reach maximum plasma concentration after dosing
Clearance rate (CL) | Within 60 minutes before administration to 1680 hours after administration.
  Percentage of the organ-scavenging drugs that eliminated by the body
Half-life (T1/2) | Within 60 minutes before administration to 1680 hours after administration.
  The time it takes for serum drug concentrations to drop by half
Apparent volume of distribution (Vd) | Within 60 minutes before administration to 1680 hours after administration.
  Apparent volume of distribution after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun, Jilin, China